CLINICAL TRIAL: NCT06984445
Title: Analysis of Cord Blood S100B Protein Levels in Neonates With Fetal Anemia Due to Hemolytic Disease Undergoing Intrauterine Transfusions: A Prospective Cohort Study
Brief Title: Cord Blood S100B Protein Levels in Neonates Following Intrauterine Transfusions for HDFN-Associated Fetal Anemia
Status: Recruiting | Type: Observational
Sponsor: Institute of Mother and Child, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Agnieszka Drozdowska-Szymczak, MD, PhD, Institute of Mother and Child, Warsaw, Poland
Other Study IDs: S100BIUT
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: s100b; Hypoxia-Ischemia, Brain; Hemolytic Disease of the Fetus and Newborn; Fetal Anemia
Keywords: S100B protein; hemolytic disease of fetus and newborn (HDFN); intrauterine transfusion (IUT); fetal anemia; newborn; central nervous system (CNS) damage; CNS hypoxia-ischemia (HI)
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Erythroblastosis, Fetal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and whole blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study group: Pregnant women with HDFN-related fetal anemia requiring intrauterine transfusion (IUT). The need for IUT is determined based on prenatal ultrasound assessment of the peak systolic velocity in the middle cerebral artery (MCA-PSV), expressed as multiples of the median (MoM). A MoM value greater than 1.5 is indicative of severe fetal anemia and serves as the primary criterion for IUT.
  Interventions: Diagnostic Test: Cord blood S100B protein level prior to IUT; Diagnostic Test: Umbilical cord blood gas analysis prior to IUT; Diagnostic Test: Fetal blood count evaluation prior to IUT; Diagnostic Test: Cord blood S100B protein concentration at birth; Diagnostic Test: Umbilical cord blood gas analysis at birth; Diagnostic Test: Complete blood count after birth; Diagnostic Test: Ultrasound evaluation of fetal blood flow; Diagnostic Test: Neonatal transfontanelle ultrasound assessment; Diagnostic Test: Complete blood count analysis in cord blood at birth
- Control group: Women with pregnancies complicated by HDFN who do not meet the criteria for intrauterine transfusion (IUT).
  Interventions: Diagnostic Test: Cord blood S100B protein concentration at birth; Diagnostic Test: Umbilical cord blood gas analysis at birth; Diagnostic Test: Complete blood count after birth; Diagnostic Test: Ultrasound evaluation of fetal blood flow; Diagnostic Test: Neonatal transfontanelle ultrasound assessment; Diagnostic Test: Complete blood count analysis in cord blood at birth

INTERVENTIONS:
Diagnostic Test: Cord blood S100B protein level prior to IUT — One milliliter of cord blood will be collected before each IUT procedure to measure S100B protein concentration. The sample will be labeled with the mother's name, date of birth, collection date, and IUT indication, then sent to the laboratory for centrifugation.
  Groups: Study group
Diagnostic Test: Umbilical cord blood gas analysis prior to IUT — Half a milliliter of cord blood will be collected before each IUT procedure for immediate umbilical cord blood gas analysis, including pH, base excess (BE), and lactate levels.
  Groups: Study group
Diagnostic Test: Fetal blood count evaluation prior to IUT — Fetal blood count data, including hemoglobin and hematocrit levels, will be collected before each IUT procedure.
  Groups: Study group
Diagnostic Test: Cord blood S100B protein concentration at birth — After delivery, one milliliter of blood will be collected from the severed umbilical cord to measure the concentration of S100B protein. The sample will be labeled with the mother's name, the child's birth date and sex, and the collection date, before being sent to the laboratory for centrifugation.
Diagnostic Test: Umbilical cord blood gas analysis at birth — After birth, 0.5 mL of blood will be collected from the severed umbilical cord to assess pH, base excess (BE), and lactate levels in an umbilical cord blood gas analysis.
Diagnostic Test: Complete blood count after birth — Complete blood count parameters, including hematocrit (Hct) and hemoglobin (Hgb) concentrations, will be measured within six hours after birth.
Diagnostic Test: Ultrasound evaluation of fetal blood flow — Fetal cerebral blood flow will be routinely assessed via ultrasound, including measurements of MCA-PSV values.
Diagnostic Test: Neonatal transfontanelle ultrasound assessment — A transfontanelle ultrasound examination will. be performed to assess for any abnormalities in the newborn.
Diagnostic Test: Complete blood count analysis in cord blood at birth — Complete blood count parameters, including hematocrit (Hct) and hemoglobin (Hgb) concentrations, will be measured in cord blood samples collected at birth.

SUMMARY:
levated levels of S100B protein are a well-established marker of central nervous system (CNS) damage. Fetal anemia resulting from hemolytic disease of the fetus and newborn (HDFN) often necessitates intrauterine transfusions (IUTs) and represents a significant risk factor for CNS injury. However, it remains uncertain whether S100B protein levels can reliably predict which fetuses are at higher risk for CNS complications in this context. Furthermore, the potential role of measuring S100B concentrations before IUT in prenatal assessments, and its relationship to the severity of anemia and fetal cerebral blood flow, remains poorly understood. This study aims to investigate the concentration of S100B protein in cord blood from newborns with HDFN-related fetal anemia requiring IUT. The study group comprises pregnancies complicated by HDFN with abnormal middle cerebral artery (MCA) blood flow, indicating the need for IUT. In this group, S100B protein levels will be measured before each IUT, with additional measurements if further transfusions are required. The control group consists of pregnancies with HDFN that do not require IUT. Cord blood samples will be collected at birth to evaluate S100B protein levels in both groups. Additionally, fetal MCA blood flow will be monitored, and in the study group, fetal hemoglobin and hematocrit levels will be assessed before each IUT. The primary endpoints of the study include the measurement of cord blood S100B protein levels before IUT in the study group and at birth in both groups. Secondary endpoints will explore the potential correlations between S100B protein levels and umbilical cord blood gas parameters (e.g., pH, BE, lactate), fetal cerebral blood flow parameters (e.g., MCA-PSV values), and blood count parameters (e.g., hemoglobin and hematocrit levels), both before IUT in the study group and after birth in both groups.

ELIGIBILITY:
Study Group - Inclusion Criteria:

1. Singleton pregnancy.
2. Diagnosis of HDFN confirmed by the detection of alloantibodies through maternal blood screening.
3. Availability of complete medical records, including routine ultrasound assessments of fetal MCA blood flow.
4. Fetal anemia requiring IUT, indicated by a MCA-PSV MoM value exceeding 1.5.

Study Group - Exclusion Criteria:

1. Maternal chronic use of selective serotonin reuptake inhibitors (SSRIs).

Control Group - Inclusion Criteria:

1. Singleton pregnancy.
2. Diagnosis of HDFN confirmed by the detection of alloantibodies through maternal blood screening.
3. Availability of complete medical records, including routine ultrasound assessments of fetal MCA blood flow.
4. No indications for IUT, as determined by MCA-PSV MoM values <1.5 in routine assessments of fetal cerebral arterial flow.

Control Group - Exclusion Criteria:

1. Maternal chronic use of selective serotonin reuptake inhibitors (SSRIs).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women diagnosed with hemolytic disease of the fetus and newborn (HDFN).
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Cord blood S100B protein concentration | Within 3 months of enrollment
  Cord blood S100B protein concentration, measured both before the IUT in the study group and from umbilical cord blood samples collected after birth in both the study and control groups.

SECONDARY OUTCOMES:
Correlation of cord blood S100B concentration with pH, BE, and lactate levels in cord blood gas analysis | Within 3 months of enrollment
  The correlation between cord blood S100B protein concentration and pH, BE, and lactate levels, measured before the IUT in the study group and from umbilical cord blood samples collected after birth in both the study and control groups.
Association between cord blood S100B protein concentration and complete blood count parameters | Within 3 months of enrollment
  The relationship between cord blood S100B protein concentration and Hgb and Hct levels, measured from cord blood samples collected before IUT in the study group, as well as from cord blood at birth and venous blood within the first six hours of life in both groups.
Correlation between cord blood S100B protein concentration and MCA-PSV values | Within 3 months of enrollment
  The association between cord blood S100B protein concentration and MCA-PSV values determined via fetal ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka A. Drozdowska-Szymczak, MD, PhD, Principal Investigator — Institute of Mother and Child in Warsaw, Poland
Locations (1):
- Institute of Mother and Child, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ree IMC, Smits-Wintjens VEHJ, van der Bom JG, van Klink JMM, Oepkes D, Lopriore E. Neonatal management and outcome in alloimmune hemolytic disease. Expert Rev Hematol. 2017 Jul;10(7):607-616. doi: 10.1080/17474086.2017.1331124. Epub 2017 Jun 5. PMID 28503958
- [Background] Lindenburg IT, Smits-Wintjens VE, van Klink JM, Verduin E, van Kamp IL, Walther FJ, Schonewille H, Doxiadis II, Kanhai HH, van Lith JM, van Zwet EW, Oepkes D, Brand A, Lopriore E; LOTUS study group. Long-term neurodevelopmental outcome after intrauterine transfusion for hemolytic disease of the fetus/newborn: the LOTUS study. Am J Obstet Gynecol. 2012 Feb;206(2):141.e1-8. doi: 10.1016/j.ajog.2011.09.024. Epub 2011 Sep 24. PMID 22030316
- [Background] Mazarico E, Llurba E, Cumplido R, Valls A, Melchor JC, Iglesias M, Cabero L, Gratacos E, Gomez-Roig MD. Neural injury markers in intrauterine growth restriction and their relation to perinatal outcomes. Pediatr Res. 2017 Sep;82(3):452-457. doi: 10.1038/pr.2017.108. Epub 2017 May 31. PMID 28426650
- [Background] Malhotra A, Ditchfield M, Fahey MC, Castillo-Melendez M, Allison BJ, Polglase GR, Wallace EM, Hodges R, Jenkin G, Miller SL. Detection and assessment of brain injury in the growth-restricted fetus and neonate. Pediatr Res. 2017 Aug;82(2):184-193. doi: 10.1038/pr.2017.37. Epub 2017 May 17. PMID 28234891
- [Background] Strzalko B, Karowicz-Bilinska A, Wyka K, Krajewski P, Kesiak M, Kociszewska-Najman B. Serum S100B Protein Concentrations in SGA/FGR newborns. Ginekol Pol. 2021 Jun 9. doi: 10.5603/GP.a2021.0119. Online ahead of print. PMID 34105746
- [Background] Zaigham M, Lundberg F, Olofsson P. Protein S100B in umbilical cord blood as a potential biomarker of hypoxic-ischemic encephalopathy in asphyxiated newborns. Early Hum Dev. 2017 Sep;112:48-53. doi: 10.1016/j.earlhumdev.2017.07.015. Epub 2017 Jul 27. PMID 28756088
- [Background] Bouvier D, Giguere Y, Pereira B, Bernard N, Marc I, Sapin V, Forest JC. Cord blood S100B: reference ranges and interest for early identification of newborns with brain injury. Clin Chem Lab Med. 2020 Jan 28;58(2):285-293. doi: 10.1515/cclm-2019-0737. PMID 31622243
- [Background] Perrone S, Grassi F, Caporilli C, Boscarino G, Carbone G, Petrolini C, Gambini LM, Di Peri A, Moretti S, Buonocore G, Esposito SMR. Brain Damage in Preterm and Full-Term Neonates: Serum Biomarkers for the Early Diagnosis and Intervention. Antioxidants (Basel). 2023 Jan 29;12(2):309. doi: 10.3390/antiox12020309. PMID 36829868
- [Background] Friel LA, Romero R, Edwin S, Nien JK, Gomez R, Chaiworapongsa T, Kusanovic JP, Tolosa JE, Hassan SS, Espinoza J. The calcium binding protein, S100B, is increased in the amniotic fluid of women with intra-amniotic infection/inflammation and preterm labor with intact or ruptured membranes. J Perinat Med. 2007;35(5):385-93. doi: 10.1515/JPM.2007.101. PMID 17624933
- [Background] Pawluski JL, Galea LA, Brain U, Papsdorf M, Oberlander TF. Neonatal S100B protein levels after prenatal exposure to selective serotonin reuptake inhibitors. Pediatrics. 2009 Oct;124(4):e662-70. doi: 10.1542/peds.2009-0442. Epub 2009 Sep 28. PMID 19786426
- [Background] Lu H, Huang W, Chen X, Wang Q, Zhang Q, Chang M. Relationship between premature brain injury and multiple biomarkers in cord blood and amniotic fluid. J Matern Fetal Neonatal Med. 2018 Nov;31(21):2898-2904. doi: 10.1080/14767058.2017.1359532. Epub 2017 Aug 3. PMID 28738706
- [Background] Chiang LM, Chen WY, Yang YC, Jeng MJ. Elevation of serum S100 protein concentration as a marker of ischemic brain damage in extremely preterm infants. J Chin Med Assoc. 2015 Oct;78(10):610-6. doi: 10.1016/j.jcma.2015.06.009. Epub 2015 Aug 15. PMID 26285828
- [Background] Florio P, Abella R, Marinoni E, Di Iorio R, Li Volti G, Galvano F, Pongiglione G, Frigiola A, Pinzauti S, Petraglia F, Gazzolo D. Biochemical markers of perinatal brain damage. Front Biosci (Schol Ed). 2010 Jan 1;2(1):47-72. doi: 10.2741/s45. PMID 20036928
- [Background] Huang RZ, Zhang YJ, Zhang JF, Su YM, Peng LQ, Ya N. Relation between prognosis and changes of MBP and S100B in premature infants with periventricular leukomalacia. Genet Mol Res. 2015 Apr 30;14(2):4338-43. doi: 10.4238/2015.April.30.6. PMID 25966206
- [Background] Niwa Y, Imai K, Kotani T, Miki R, Nakano T, Ushida T, Moriyama Y, Kikkawa F. Relationship between cytokine profiles of cord blood and cord S100B levels in preterm infants. Early Hum Dev. 2019 Feb;129:65-70. doi: 10.1016/j.earlhumdev.2019.01.013. Epub 2019 Jan 23. No abstract available. PMID 30684905
- [Background] Metallinou D, Karampas G, Lazarou E, Iacovidou N, Pervanidou P, Lykeridou K, Mastorakos G, Rizos D. Serum Activin A as Brain Injury Biomarker in the First Three Days of Life. A Prospective Case-Control Longitudinal Study in Human Premature Neonates. Brain Sci. 2021 Sep 20;11(9):1243. doi: 10.3390/brainsci11091243. PMID 34573263
- [Background] Wirds JW, Duyn AE, Geraerts SD, Preijer E, Van Diemen-Steenvoorde JA, Van Leeuwen JH, Haas FJ, Gerritsen WB, De Boer A, Leusink JA. S100 protein content of umbilical cord blood in healthy newborns in relation to mode of delivery. Arch Dis Child Fetal Neonatal Ed. 2003 Jan;88(1):F67-9. doi: 10.1136/fn.88.1.f67. PMID 12496231
- [Background] Velipasaoglu M, Yurdakok M, Ozyuncu O, Portakal O, Deren O. Neural injury markers to predict neonatal complications in intrauterine growth restriction. J Obstet Gynaecol. 2015;35(6):555-60. doi: 10.3109/01443615.2014.978848. Epub 2014 Nov 13. PMID 25392968
- [Background] Gazzolo D, Abella R, Marinoni E, di Iorio R, Li Volti G, Galvano F, Frigiola A, Temporini F, Moresco L, Colivicchi M, Sabatini M, Ricotti A, Strozzi MC, Crivelli S, Risso FM, Sannia A, Florio P. New markers of neonatal neurology. J Matern Fetal Neonatal Med. 2009;22 Suppl 3:57-61. doi: 10.1080/14767050903181468. PMID 19718579
- [Background] Masaoka N, Nakajima Y, Morooka M, Tashiro H, Wada M, Maruta K, Iwane E, Yamashiro M. The impact of intrauterine infection on fetal brain damage assessed by S100B protein concentrations in umbilical cord arteries. J Matern Fetal Neonatal Med. 2016;29(15):2464-9. doi: 10.3109/14767058.2015.1087501. Epub 2015 Sep 30. PMID 26421445
- [Background] Debska M, Kretowicz P, Tarasiuk A, Dangel J, Debski R. Successful intrauterine treatment and good long-term outcome in an extremely severe case of fetal hemolytic disease. J Ultrason. 2014 Jun;14(57):217-22. doi: 10.15557/JoU.2014.0021. Epub 2014 Jun 30. PMID 26673879
- [Background] Fenton TR, Kim JH. A systematic review and meta-analysis to revise the Fenton growth chart for preterm infants. BMC Pediatr. 2013 Apr 20;13:59. doi: 10.1186/1471-2431-13-59. PMID 23601190
- [Background] Kwiatkowski S, Torbe A, Borowski D, Breborowicz G, Czajkowski K, Huras H, Kajdy A, Kalinka J, Kosinska-Kaczynska K, Leszczynska-Gorzelak B, Rokita W, Ropacka-Lesiak M, Sieroszewski P, Wielgos M, Zimmer M. Polish Society of Gynecologists and Obstetricians Recommendations on diagnosis and management of fetal growth restriction. Ginekol Pol. 2020;91(10):634-643. doi: 10.5603/GP.2020.0158. No abstract available. PMID 33184833
- [Background] Andrei C, Vladareanu R. The value of reference ranges for middle cerebral artery peak systolic velocity in the management of rhesus alloimmunized pregnancies. Maedica (Bucur). 2012 Jan;7(1):14-9. PMID 23118814
- [Background] Drozdowska-Szymczak A, Proczka J, Chrzanowska-Liszewska D, Truszkowski K, Mazanowska N, Krajewski P. Liver Dysfunction with Severe Cholestasis and Coagulation Disorders in the Course of Hemolytic Disease of the Newborn Requiring Chelation Therapy-A Case Report and Review of the Literature. J Clin Med. 2023 Dec 13;12(24):7645. doi: 10.3390/jcm12247645. PMID 38137714
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. BMJ. 2007 Oct 20;335(7624):806-8. doi: 10.1136/bmj.39335.541782.AD. PMID 17947786
- [Background] Cuschieri S. The STROBE guidelines. Saudi J Anaesth. 2019 Apr;13(Suppl 1):S31-S34. doi: 10.4103/sja.SJA_543_18. PMID 30930717
- [Background] Gordijn SJ, Beune IM, Thilaganathan B, Papageorghiou A, Baschat AA, Baker PN, Silver RM, Wynia K, Ganzevoort W. Consensus definition of fetal growth restriction: a Delphi procedure. Ultrasound Obstet Gynecol. 2016 Sep;48(3):333-9. doi: 10.1002/uog.15884. PMID 26909664
- [Background] Society for Maternal-Fetal Medicine (SMFM). Electronic address: pubs@smfm.org; Mari G, Norton ME, Stone J, Berghella V, Sciscione AC, Tate D, Schenone MH. Society for Maternal-Fetal Medicine (SMFM) Clinical Guideline #8: the fetus at risk for anemia--diagnosis and management. Am J Obstet Gynecol. 2015 Jun;212(6):697-710. doi: 10.1016/j.ajog.2015.01.059. Epub 2015 Mar 27. PMID 25824811
- [Background] Jung E, Romero R, Suksai M, Gotsch F, Chaemsaithong P, Erez O, Conde-Agudelo A, Gomez-Lopez N, Berry SM, Meyyazhagan A, Yoon BH. Clinical chorioamnionitis at term: definition, pathogenesis, microbiology, diagnosis, and treatment. Am J Obstet Gynecol. 2024 Mar;230(3S):S807-S840. doi: 10.1016/j.ajog.2023.02.002. Epub 2023 Mar 21. PMID 38233317